CLINICAL TRIAL: NCT06702423
Title: Enhancing Health Literacy Through Artificial Intelligence-Powered Chatbot: a Randomized Controlled Trial on Addressing Human Papillomavirus Vaccination Misinformation Among Caregivers in Japan
Brief Title: Enhancing Health Literacy Through AI-Powered Chatbot: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Nagasaki University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UW231392; NCT06718166 (obsolete NCT alias)
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: HPV vaccine; AI; chatbot; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-based chatbot (Experimental): A chatbot that was developed using information related to HPV vaccines from authoritative sources such as the Japanese Ministry of Health, Labour, and Welfare, World Health Organization, Centers for Disease Control and Prevention, and other reputable public health organizations and validated survey questions from published research.
  Interventions: Behavioral: AI-based chatbot
- Leaflet (Active Comparator): A leaflet which is a publicly accessible HPV vaccination document prepared by the Ministry of Health, Labour, and Welfare.
  Interventions: Behavioral: Leaflet

INTERVENTIONS:
Behavioral: AI-based chatbot — A tailored Japanese HPV vaccination chatbot.
  Arms: AI-based chatbot
Behavioral: Leaflet — A publicly accessible HPV vaccination leaflet prepared by the Ministry of Health, Labour, and Welfare.
  Arms: Leaflet

SUMMARY:
The goal of this study is to learn if an innovative digital artificial intelligence (AI)-based communication tool works to enhance health literacy among Japanese caregivers regarding Human Papillomavirus (HPV) vaccination.

Participants will:

* Answer a pre-intervention survey, get information regarding HPV vaccination from an AI-based chatbot or leaflet, and answer a post-intervention survey.
* Continue interacting with the chatbot or leaflet for two weeks.
* Answer a follow-up survey.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and feasibility of an AI-driven chatbot in enhancing caregivers' health literacy about HPV vaccination and examines its impact on informed decision-making concerning their daughters' vaccination through a randomized controlled trial (RCT). To achieve this, the study will undertake the following interconnected activities:

1. Randomized Controlled Trial Participants will be randomly assigned to either the control or intervention group. Those in the control group will spend 5-10 minutes reading a publicly accessible HPV vaccination leaflet prepared by the MHLW, serving as the standard of care. Conversely, participants in the intervention group will be invited to interact with the chatbot for 5-10 minutes, posing inquiries (n>10) about HPV vaccination policies and related topics in Japan. Pre- and post-intervention assessments, as detailed below, will be administered to evaluate the chatbot's effectiveness and feasibility to counter HPV vaccine misinformation and support caregivers' vaccination decision-making processes.
2. Pre- and post-intervention assessments Following informed consent and enrollment, participants will complete a pre-intervention survey to establish baseline data. Post-intervention survey will be introduced at two touchpoints: the first is directly after spending time with either a leaflet (control) or a chatbot (intervention), and the second is two weeks after the first touchpoint.

The surveys are designed to assess the chatbot's effectiveness in enhancing caregivers' digital health literacy about HPV vaccination and facilitating informed vaccine decision-making.

ELIGIBILITY:
Inclusion Criteria:

* A nationally representative sample of female caregivers with daughters aged 12-18 who have not received any HPV vaccine.
* Those who have access to a smartphone or computer with internet connectivity to interact with experiment materials (chatbot or online leaflet).
* Those who provide informed consent and agree to participate in the study.

Exclusion Criteria:

* Those who need help reading through the participant information sheet, providing consent online, accessing experiment materials (chatbot or online leaflet), or answering surveys will be excluded. This may include people who do not have access to an online environment or people with severe cognitive impairments who cannot interact with the experiment materials. Also, those who have participated or are participating in similar studies regarding vaccination or experiments that utilize chatbots will be excluded.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 844 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
health literacy | 2 weeks
  Health literacy related to HPV vaccination will be measured by changes in caregivers' scores on questions concerning facts about HPV vaccines and associated health information. This metric will be evaluated by determining the proportion of respondents who correctly answer these questions, reflecting their understanding and knowledge.

SECONDARY OUTCOMES:
decision-making | 2 weeks
  Decision-making regarding HPV vaccination will be evaluated based on changes in the uptake status of HPV vaccines among caregivers' daughters. This will be measured by the proportion of respondents who answer 'Yes' to the question, 'Have you decided to vaccinate your daughter against HPV?' Response options will include 'Yes' and 'No.'

CONTACTS AND LOCATIONS:
Overall Officials: Leesa Lin, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom